CLINICAL TRIAL: NCT01411007
Title: The Impact of Real-time fMRI Feedback on Response to Nicotine Cues
Brief Title: The Impact of Real-time Functional Magnetic Resonance Imaging (fMRI) Feedback on Response to Nicotine Cues
Acronym: RTSmoking
Status: Terminated | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: HR#19231
Record Dates: First submitted 2011-08-04; First posted 2011-08-05 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2011-07

CONDITIONS: Nicotine Dependence
Keywords: Nicotine; Cigarettes; Smoker; realtime fMRI; brain imaging; imaging
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Smokers: Nicotine addicted smokers, smoking an average of at least 10 cigarettes per day.
- Non-Smokers

SUMMARY:
The purpose of this study is to develop a technique to provide feedback of brain activity and to use this technique to reduce levels of craving in nicotine dependent smokers. The researchers will use a brain scan called functional magnetic resonance imaging (MRI). MRI uses magnets to take pictures of your brain. Functional MRI measures brain blood flow that is related to brain activity. This measure of brain activity can be presented or "feedback" to volunteers.

DETAILED DESCRIPTION:
There are three total visits for this study. Details of each visit are listed below.

Screening/Assessment Visit:

This evaluation will include interviews, questionnaires, computerized testing, urine drug screen, breath sample for carbon monoxide level and alcohol and physical examination. If accepted into this study, you will then be scheduled for a biofeedback and an imaging session. Both smokers and nonsmoking controls will go through the screening process.

Biofeedback Session:

You will be asked to participate in a biofeedback session scheduled for 60 minutes. You will be comfortably seated and a sensor to measure your temperature will be placed on a finger of your non-dominant hand. You will be asked to make changes in your skin temperature based on feedback from the monitoring system. Your responses to the biofeedback session will be compared to your responses to feedback in the scanner. Both smokers and nonsmoking controls will go through the biofeedback session.

Imaging Visit:

The imaging visit should last approximately 2 hours. You will also be asked to refrain from using alcohol and any street drugs for 24 hours and from using any marijuana for 3 days prior to the visit. If you smoke, you will be asked not to smoke for 2 hours prior to the scanning session. Evaluation will include an interview, questionnaires, and a breath carbon monoxide level. If you are a woman, a urine pregnancy test will be completed prior to the exam. If you smoke, you will be asked to complete questionnaires that focus on your craving and withdrawal symptoms for cigarettes. These questionnaires will take approximately 15 minutes to complete.

ELIGIBILITY:
Inclusion Criteria (all participants):

1. Age 18 - 60 right handed adults.
2. General good health confirmed by history & physical.
3. Able to read and understand questionnaires and informed consent.
4. Participants must have a negative urine drug screen (UDS) and pregnancy test prior to imaging sessions.
5. Female participants will use a reliable method of birth control throughout the study.

Additional Inclusion Criteria for non-smoking group:

1. Has used tobacco products no more than on experimental basis (none in past year).

Additional Inclusion Criteria for smoking group:

1. Smokers must meet criteria for primary nicotine dependence confirmed by Fagerström Test for Nicotine Dependence (FTND) and smoking on average 10 cigarettes a day in the last 30 days prior to assessment.
2. Smokers must be motivated to quit.
3. Demonstrate subjective craving as measured by the Questionnaire of Smoking Urges (QSU)-B.

Exclusion Criteria:(all participants):

1. Meets the Diagnostic and Statistical Manual (DSM)-IV criterion for lifetime or current substance dependence except for nicotine dependence.
2. Any psychoactive substance abuse within the last 30 days as evidenced by subject report or urine drug screen.
3. Use of other tobacco products.
4. Current use of nicotine replacement therapy, bupropion, varenicline, or other smoking cessation treatment.
5. Healthy volunteers must not have had more than experimental use of cigarettes.
6. Meets DSM-IV criteria for current axis I disorders of major depression, panic disorder, obsessive compulsive disorder, post-traumatic stress syndrome, bipolar affective disorder, schizophrenia, or any other psychotic disorder or organic mental disorder. The rationale for excluding them is that symptoms from these disorders may affect dependent variables and complicate interpretation of the data.
7. Current suicidal ideation with plan or homicidal ideation.
8. Need for maintenance or acute treatment with any psychoactive medication including anti-seizure medications which could potentially interfere with fMRI.
9. Clinically significant medical problems that would impair participation or limit ability to participate in scan.
10. Sexually active females of child-bearing potential who are pregnant (by urine HCG), nursing, or who are not using a reliable form of birth control.
11. Has current charges pending for a violent crime (not including Driving Under the Influence (DUI) related offenses).
12. Persons with ferrous metal implants or pacemaker since fMRI will be used.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult nicotine dependant smokers and Healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2010-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S George, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States